CLINICAL TRIAL: NCT00247585
Title: Hangover, Congeners, Sleep and Occupational Performance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NIAAAHOW12087; NIH Grant R01 AA12087-04A1
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2006-12-06 (Estimated); Status verified 2006-12

CONDITIONS: Sleep; Neurobehavioral Manifestations
Keywords: Alcohol; Alcohol abuse; Alcohol consumption; Unhealthy alcohol use; Residual effects; Sleep Stages; Respiratory Physiology
MeSH Terms: conditions — Neurobehavioral Manifestations; Alcoholism; Alcohol Drinking | interventions — Ethanol

INTERVENTIONS:
Drug: Ethanol (Bourbon or Vodka)

SUMMARY:
The objective is to investigate residual effects of heavy drinking, with or without hangover symptoms. The primary aim is to test several hypotheses about residual effects of heavy drinking. Hypotheses about how heavy drinking affects next-day performance include direct physiological effects of alcohol, alcohol withdrawal effects, and non-ethanol effects, such as congeners, or family history of alcohol problems. The investigators will test the following hypotheses:

1. relative to placebo, heavy drinking will degrade next-day performance, and this relationship will be mediated in full or in part by quality of sleep;
2. a high congener alcoholic beverage will affect performance to a greater degree than a low congener beverage and this relationship will be mediated by severity of hangover symptoms.

DETAILED DESCRIPTION:
The primary aim of the proposed study is to test several hypotheses about residual effects of heavy drinking. Hypotheses about how heavy drinking affects next-day performance include direct physiological effects of alcohol (e.g., electrolyte imbalance, low blood sugar, sleep disturbance), alcohol withdrawal effects, acetaldehyde toxicity, and non-ethanol effects, such as congeners or family history of alcohol (Swift and Davidson, 1998). Using a placebo-controlled randomized trial, we will dose participants with placebo or with a high or low congener alcoholic beverage (to a level of 0.10 g% BAC) the night before they perform exercises on a neurobehavioral evaluation system. We will monitor participants' sleep to assess sleep disturbance. We will collect information on hangover symptoms the morning after dosing. We will also collect data on participants' family history of drinking problems. We will test the following hypotheses:

1. relative to placebo, heavy drinking will degrade next-day cognitive performance, and this relationship will be mediated in full or in part by quality of sleep; and
2. a high congener alcoholic beverage will affect performance to a greater degree than a low congener beverage and this relationship will be mediated by severity of hangover symptoms.

We will explore whether the residual effects of heavy drinking on next-day cognitive performance are attenuated among participants positive for a family history of alcohol problems, relative to family-history-negative participants.

A secondary aim is to test the effectiveness of the Psychomotor Vigilance Test (PVT), a validated measure of fatigue, as a fitness-for-duty test. We will test whether the PVT can distinguish dosing status (alcohol or placebo) of participants at the time performance is measured the next day and the extent to which PVT measures correlate with performance scores.

Participants will be young adults ages 21-30 who are currently enrolled in an undergraduate college or university or have graduated from a college or university. Alcoholic beverages will be bourbon (high-congener) in soda or vodka (low-congener) in soda. Placebo will be tonic alone. We will use a mixed within- and between-subjects design, balancing the order of placebo and alcohol administration. Performance will be measured using a computer-based neurobehavioral evaluation system.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-30
* Currently enrolled or have completed college/university
* Have had 5 or more drinks (4 if female) in the last 30 days
* Score less than a 5 on the Short Michigan Alcohol Screening Test (SMAST)
* No self-reported history of counseling or treatment for substance abuse
* Not taking any medication contraindicated for alcohol use or that disrupts sleep
* Doesn't have a health condition contraindicated for alcohol use
* Has not been diagnosed with a primary sleep disorder
* Has not been diagnosed with a mental health disorder
* Not currently working night shifts at a job
* Not routinely taking medications that affect sleep
* No evidence of extreme morningness or eveningness as assessed by questionnaire
* Not a regular smoker

Exclusion Criteria:

* Less than age 21 and greater than age 30
* Not currently enrolled or has not completed college/university
* Hasn't had 5 or more drinks (4 if female) in the last 30 days (not a regular drinker)
* Score greater than or equal to 5 on the Short Michigan Alcohol Screening Test (SMAST)
* Self-reported history of counseling or treatment for substance abuse
* Taking any medication contraindicated for alcohol use or that disrupts sleep
* Has a health condition contraindicated for alcohol use
* Has been diagnosed with a primary sleep disorder
* Has been diagnosed with a mental health disorder
* Currently working night shifts at a job
* Routinely taking medications that affect sleep
* Evidence of extreme morningness or eveningness as assessed by questionnaire
* Is a regular smoker
* Not a regular drinker
* Is pregnant or nursing

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140
Dates: Start 2003-09; Study Completion 2006-06

PRIMARY OUTCOMES:
Cognitive function in response to heavy drinking
Cognitive function in response to sleep quality
Self-reported residual effects of heavy drinking

SECONDARY OUTCOMES:
Effectiveness of psychomotor vigilance testing as a fitness-for-duty test

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Howland, PhD, MPH, MPA, Principal Investigator — Boston University
Locations (1):
- General Clinical Research Center, Boston University School of Public Health/Boston Medical Center, Boston, Massachusetts, United States